CLINICAL TRIAL: NCT00406406
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SKI-606 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating SKI-606 Administered to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3160A1-103
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — bosutinib

INTERVENTIONS:
Drug: SKI-606

SUMMARY:
Safety and tolerability of SKI-606 in healthy subjects; the influence of food intake on the same.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics; safety and tolerability; influence of food.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com
Locations (1):
- Utrecht, Netherlands